CLINICAL TRIAL: NCT02685046
Title: Targeted Therapy With Imatinib for Treatment of Poor Prognosis Mesenchymal-type Resectable Colon Cancer: a Proof-of-concept Study in the Preoperative Window Period.
Brief Title: Imatinib as Pre-operative Anti-Colon Cancer Targeted Therapy
Acronym: ImPACCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: UMC Utrecht (Other)
Collaborators: Meander Medical Center (Other); Erasmus Medical Center (Other); Hubrecht Institute (Unknown)
Responsible Party: Principal Investigator, Prof dr I.H.M. Borel Rinkes, Chief Surgical Specialities, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-TT-IMA-14; NL50620.041.15 (Registry Identifier: CCMO); 2014-003965-11 (EudraCT Number)
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Subjects will be treated with the medicinal product imatinib, which will be administered orally in tablets of 400mg, once per day, during two weeks prior to tumor resection.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Subjects will be treated with the medicinal product imatinib, which will be administered orally in tablets of 400mg, once per day, during two weeks prior to tumor resection.
  Other Names: Gleevec; STI571

SUMMARY:
In this proof-of-concept trial the investigators will study the effects of imatinib treatment on the biology of mesenchymal-type colon cancers.

DETAILED DESCRIPTION:
Tumor biopsies from patients with newly diagnosed colon cancer will be pre-screened with an RT-qPCR test to identify tumors of the mesenchymal subtype. Patients with mesenchymal-type tumors that meet the in- and exclusion criteria will be treated with imatinib during the "window period" that normally precedes surgery. Immediately following tumor resection, biopsies will be taken from the surgical specimen. Gene and protein expression of the pre- and post-treatments biopsies will be compared to assess the effects of imatinib therapy on PDGFR- and cKIT-signalling and on the mesenchymal gene expression profile.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years
2. Histologically proven adenocarcinoma of the colon;
3. Completed cancer staging with CT-abdomen and CT-thorax/X-thorax according to hospital's standard of care;
4. Confirmed eligibility for surgery with curative intent as deemed by the hospital's multidisciplinary board (MDB) review;
5. An intratumoural gene expression profile of PDGFR-α, PDGFR-β, PDGF-C and KIT, indicative of the mesenchymal phenotype, according to our diagnostic RT-qPCR test (i.e. more than 50% chance of having the mesenchymal phenotype);
6. Minimum of four properly stored pre-treatment biopsies for gene expression analysis/ELISA;
7. WHO performance status 0 or 1;
8. Adequate haematology status and organ function, defined as:

   * Normal creatinine clearance (≥60 ml/min (MRDR))
   * ALAT within 2.5x upper limit of normal (ULN)
   * PT-INR < 1.5
   * Leukocytes > 1,5*10^9/L; Hb > 6.0 mmol/L; platelets > 100*10^9/L
9. Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests;
10. Written informed consent.

Exclusion Criteria:

1. The presence of synchronous distant metastases;
2. Current hospital standard of care dictates that subject should undergo any neoadjuvant therapy;
3. Concurrent participation in another clinical trial using any medicinal product, or participation in such a trial in the period of three months prior to the current trial;
4. Women who are pregnant, plan to become pregnant or are lactating during the study or for up to 30 days after the last dose of imatinib;
5. Known HIV or Hepatitis B/C infection;
6. Known symptomatic congestive heart failure;
7. Co-morbidity requiring concomitant treatment with drugs that act as strong inducers of CYP3A4 or with drugs with a narrow therapeutic range influenced by imatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04; Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Effects of treatment on the mesenchymal gene expression profile | period from diagnostic colonoscopy until surgical resection (~5 weeks)
  To assess the extent of change in the mesenchymal phenotype, gene expression arrays will be generated from pre- and post-treatment tissue samples and the expression of genes associated with the poor-prognosis mesenchymal subtype will be compared.

SECONDARY OUTCOMES:
Extent of targeted inhibition of PDGFR and KIT phosphorylation in cancer cells | period from diagnostic colonoscopy until surgical resection (~5 weeks)
  I. Measurement of PDGFR and cKIT inhibition by comparison of the fraction of autophosphorylated PDGFR and cKIT pre-treatment versus post-treatment, measured with ELISA on tissue samples derived from diagnostic biopsies and surgery.
Correlation between plasma imatinib trough levels on day 14 and intratumoural concentration of imatinib in the resection specimen | at time of surgery
Correlation between the extent of PDGFR and cKIT inhibition and systemic and intratumoural imatinib and CGP74588 concentration | at time of surgery
Change in plasma CEA-concentrations | period between diagnostic colonoscopy until surgical resection (~5 weeks)
Change in plasma levels of circulating tumor DNA | period between diagnostic colonoscopy until surgical resection (~5 weeks)
Effects of imatinib on the ability of cancer cells to form in vitro 3D cell cultures (organoids) | at time of surgery
  V. The ability to establish organoids from imatinib-treated tumours will be compared with the general success rate of organoid formation from colon tumours at the Hubrecht Institute.
Number of participants with treatment-related adverse events as assessed by CTCAEv4.02 | from start of treatment until 2 weeks after last dose imatinib
  The occurrence, frequency and severity of adverse events during preoperative treatment with imatinib, peroperatively or in the postoperative period (up to 14 days after tumour resection).

CONTACTS AND LOCATIONS:
Overall Officials: I HM Borel Rinkes, MD, PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Netherlands (3):
  - Meander Medical Center, Amersfoort, Utrecht
  - Diakonessenhuis, Utrecht
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ubink I, Bloemendal HJ, Elias SG, Brink MA, Schwartz MP, Holierhoek YCW, Verheijen PM, Boerman AW, Mathijssen RHJ, de Leng WWJ, de Weger RA, van Grevenstein WMU, Koopman M, Lolkema MP, Kranenburg O, Borel Rinkes IHM. Imatinib treatment of poor prognosis mesenchymal-type primary colon cancer: a proof-of-concept study in the preoperative window period (ImPACCT). BMC Cancer. 2017 Apr 19;17(1):282. doi: 10.1186/s12885-017-3264-y. PMID 28424071